CLINICAL TRIAL: NCT03525756
Title: Cystogram for Early Foley Catheter Removal Post Colovesical Fistula Resection
Brief Title: Cystogram Before Removal of Foley Catheter After Repair of Colovesical Fistula
Status: Completed | Type: Observational
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 171002-1
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Colovesical Fistula
Keywords: cystogram; Foley catheter
MeSH Terms: conditions — Intestinal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystogram on Post-Op Day 2: An indwelling Foley catheter is placed intraoperative and continued postoperative. All patients who consent to participate would undergo a cystogram on postoperative day two. The cystogram will be conducted by a radiologist and technician well-trained in the techniques and interpretation of the study. The colorectal surgery enhanced recovery protocol will be followed on all patients with the exception of the cystogram being conducted on post-op day two.

SUMMARY:
Colovesical fistulas are well-recognized but relatively uncommon pathology to both the general and colorectal surgeon. It is a complication arising from an underlying primary acute to chronic inflammatory process. Although colovesical fistulas are uncommon, they are associated with significant morbidity, affect quality of life, and may lead to death, usually secondary to urosepsis. Early diagnosis and management is essential.

The purpose of the study is to determine the objective use of cystographic evaluation on postoperative day two to guide early Foley catheter removal post colovesical fistula takedown. The hypothesis is that a cystogram showing no extravasation of contrast on postoperative day two will predict safe removal without increased morbidity.

This is an uncontrolled, single arm trial. Patients who meet criteria to undergo either minimally invasive or open colovesical fistula takedown with sigmoid colectomy, without evidence of the need for bladder repair will be eligible to participate. An indwelling Foley catheter is placed intraoperative and continued postoperative. All patients who consent to participate would undergo a cystogram on postoperative day two. The cystogram will be conducted by a radiologist and technician well-trained in the techniques and interpretation of the study. The colorectal surgery enhanced recovery protocol will be followed on all patients with the exception of the cystogram being conducted on post-op day two. If there is no evidence of extravasation of dye is seen on the cystogram the Foley catheter will be removed. Patients will be monitored closely following catheter removal to ensure self-diuresis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with clinical, radiographic, or endoscopic confirmation of a colovesical fistula
* patients undergoing either minimally invasive or open colovesical fistula takedown with sigmoid colectomy, without evidence of the need for bladder repair

Exclusion Criteria:

* malignant disease
* Crohn's disease
* radiation-induced colovesical fistula
* current pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting all inclusion and no exclusion criteria being cared for at Mount Carmel Health System
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Successful Foley Catheter Removal at Day 2 | 16 Hours After Foley Catheter Removal
  Defined as no evidence of extravasation of dye is seen on the cystogram on day two, followed by successful self diuresis within 16 hours of Foley catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Jaswant Madhavan, MD, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States